CLINICAL TRIAL: NCT03976713
Title: Bufei Yishen Granule for Reducing Acute Exacerbation in GOLD Stage 3 or 4 COPD: A Randomized, Double-blind, Placebo Controlled Trial
Brief Title: Bufei Yishen Granule for Reducing Acute Exacerbation in GOLD Stage 3 or 4 COPD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Collaborators: ShuGuang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCM for GOLD stage 3 or 4 COPD
Record Dates: First submitted 2019-05-29; First posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Bufei Yishen Granule; Randomized Controlled Trial
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bufei Yishen granule plus Western medicine (Experimental): Patients in this arm will receive Bufei Yishen granule in addition to Western medicine.
  Interventions: Drug: Bufei Yishen granule; Drug: Tiotropium Bromide Powder for Inhalation
- Placebo Bufei Yishen granule plus Western medicine (Placebo Comparator): Patients in this arm will receive placebo Bufei Yishen granule in addition to Western medicine.
  Interventions: Drug: Placebo Bufei Yishen granule; Drug: Tiotropium Bromide Powder for Inhalation

INTERVENTIONS:
Drug: Bufei Yishen granule — Bufei Yishen granule will be administered twice daily for five days a week for 52 weeks.
  Arms: Bufei Yishen granule plus Western medicine
Drug: Placebo Bufei Yishen granule — Placebo Bufei Yishen granule will be administered twice daily for five days a week for 52 weeks. The placebo granule consists of dextrin, bitter and 5% of the Bufei Yishen granule. The appearance, weight, color and odor of the preparation are the same as those of treatment group.
  Arms: Placebo Bufei Yishen granule plus Western medicine
Drug: Tiotropium Bromide Powder for Inhalation — Tiotropium Bromide Powder for Inhalation will be used once daily (18 μg each time) for 52 weeks.

SUMMARY:
This study aims to establish the treatment scheme of Bufei Yishen granule for GOLD stage 3 or 4 chronic obstructive pulmonary disease (COPD), reducing acute exacerbation, improving exercise capacity and forming high quality evidence.

DETAILED DESCRIPTION:
COPD is a highly prevalent disease, with a prevalence among people 40 years of age or older of 10.1% worldwide and 13.7% in China. COPD has become the third leading cause of death worldwide. Frequent acute exacerbation and exercise limitation broadly exist in COPD patients, especially those in GOLD stage 3 or 4. Although appropriate pharmacological therapies have been proven to be effective in COPD management, however, many gaps are still to be filled. For example, the adverse effects of pharmacologic therapies can never be ignored. The investigator's previous studies suggested that traditional Chinese medicine (TCM) has effect on GOLD stage 3 or 4 COPD.

This is a multicenter, randomized, double-blind, placebo controlled trial to evaluate the effect of Bufei Yishen granule on reducing acute exacerbation in GOLD stage 3 or 4 COPD subjects. After a 14-day run-in period, 348 subjects will be randomly assigned to treatment group or control group for 52-week treatment. The primary outcomes are frequency and duration of acute exacerbation. The secondary outcomes include mortality, pulmonary function, clinical symptoms, exercise capacity, quality of life and treatment satisfaction. Safety will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of GOLD stage 3 or 4 COPD.
* Syndrome differentiation meets criteria of Qi deficiency of the lung and spleen syndrome, Qi deficiency of the lung and kidney syndrome or Qi and Yin deficiency of the lung and kidney syndrome.
* Age ranges from 40 years to 80 years.
* With informed consent signed.

Exclusion Criteria:

* Pregnant and lactating women.
* Patients with severe cardiovascular and cerebrovascular diseases.
* Patients with severe liver and kidney diseases.
* Patients with asthma, bronchiectasis, active pulmonary tuberculosis, pulmonary embolism, chronic respiratory failure or other severe respiratory diseases.
* Patients with tumor after resection, radiotherapy or chemotherapy in the past 5 years.
* Patients with severe neuromuscular disorders, severe arthritis or severe peripheral vascular diseases.
* Patients with severe cognitive and psychiatric disorders.
* Patients with diabetes.
* Patients who were administered oral glucocorticoids in the past 4 weeks.
* Patients who have participated in other clinical studies in the past 4 weeks.
* People who are allergic to the treatment drugs.
* Patients who have experienced one or more acute exacerbation in the past 4 weeks.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of acute exacerbation | Up to week 52.
  Frequency of acute exacerbation will be recorded.
Duration of acute exacerbation | Up to week 52.
  Duration of acute exacerbation will be recorded.

SECONDARY OUTCOMES:
Mortality | Up to week 52.
  The mortality will be calculated.
FEV1 | Change from baseline FEV1 at week 26 and 52.
  Forced expiratory volume in one second ( FEV1) will be used to assess pulmonary function.
Clinical symptom assessment questionnaire | Change from baseline clinical symptom assessment questionnaire scores at week 13, 26, 39 and 52.
  Clinical symptom assessment questionnaire of COPD will be used to assess symptom.
6MWD | Change from baseline 6MWD at week 13, 26, 39 and 52.
  Six-minute walk distance (6MWD) will be conducted to assess exercise capacity
CAT | Change from baseline CAT scores at week 13, 26, 39 and 52.
  COPD assessment test (CAT) will be used to assess quality of life.
SF-36 | Change from baseline SF-36 scores at week 13, 26, 39 and 52.
  The MOS 36-Item Short-Form Health Survey (SF-36) will be used to assess quality of life.
mCOPD-PRO | Change from baseline mCOPD-PRO scores at week 13, 26, 39 and 52.
  The modified COPD patient-reported outcome scale (mCOPD-PRO) will be used to assess quality of life. The mCOPD-PRO contains 27 items in three domains. mCOPD-PRO scores range from 0 to 4 with a decrease in score showing higher health status.
mESQ-COPD | Change from baseline mESQ-COPD scores at week 13, 26, 39 and 52.
  The modified effectiveness satisfaction questionnaire for COPD (mESQ-COPD) will be used to assess treatment satisfaction. The mESQ-COPD contains 19 items in four domains. mESQ-COPD scores range from 0 to 4 with a decrease in score showing higher treatment satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Jiansheng Li, Professor, Study Chair — The First Affiliated Hospital of Henan University of Traditional Chinese Medicine
Locations (1):
- The First Affiliated Hospital of Henan University of Traditional Chinese Medicine, Zhengzhou, Henan, China

REFERENCES:
- [Derived] Yu XQ, Di JQ, Zhang W, Wei GS, Ma ZP, Wu L, Yu XF, Zhu HZ, Zhou M, Feng CL, Feng JH, Fan P, Li JS, Yang JY. Bu-Fei Yi-Shen Granules Reduce Acute Exacerbations in Patients with GOLD 3-4 COPD: A Randomized Controlled Trial. Int J Chron Obstruct Pulmon Dis. 2023 Nov 6;18:2439-2456. doi: 10.2147/COPD.S413754. eCollection 2023. PMID 37955027